CLINICAL TRIAL: NCT05007366
Title: Optimizing Gait Biomechanics for Posttraumatic Osteoarthritis Prevention
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: Arthritis Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Prevention
Other Study IDs: 21-1489a
Record Dates: First submitted 2021-08-12; First posted 2021-08-16 (Actual); Last update posted 2023-04-18 (Actual); Status verified 2023-04

CONDITIONS: Anterior Cruciate Ligament Injuries; Post-traumatic Osteoarthritis; Knee Osteoarthritis; Knee Injuries; Cartilage, Articular; Gait
Keywords: Biofeedback
MeSH Terms: conditions — Anterior Cruciate Ligament Injuries; Osteoarthritis, Knee; Knee Injuries

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Real-time gait biofeedback (RTGBF) (Active Comparator): The RTGBF regimen delivers biofeedback that cues a personalized target to normalize vertical ground reaction force (vGRF) of each limb.
  Interventions: Behavioral: Real-time gait biofeedback
- Sham real-time gait biofeedback (Sham RTGBF) (Sham Comparator): The Sham RTGBF regimen will receive biofeedback that cues their habitual step length determined during the accommodation period on the first session of treadmill walking.
  Interventions: Behavioral: Sham real-time gait biofeedback

INTERVENTIONS:
Behavioral: Real-time gait biofeedback — The RTGBF interventions will include eighteen step gait training sessions. The intervention will gradually increase to 3,000 steps at the 9th and 10th session with 100% feedback. During the remaining sessions, the intervention will include 3,000 steps, but the feedback will be gradually tapered off starting with the 11th session.
  Arms: Real-time gait biofeedback (RTGBF)
Behavioral: Sham real-time gait biofeedback — The Sham RTGBF interventions will include eighteen step gait training sessions. The intervention will gradually increase to 3,000 steps at the 9th and 10th session with 100% feedback. During the remaining sessions, the intervention will include 3,000 steps, but the feedback will be gradually tapered off starting with the 11th session.
  Arms: Sham real-time gait biofeedback (Sham RTGBF)

SUMMARY:
The purpose of this study is to report the feasibility and determine the initial effects of 18 sessions of real-time gait biofeedback delivered over a 6-week period on retention and transfer of normalized gait biomechanics and improvements in indicators of early post-traumatic osteoarthritis development in those with an anterior cruciate ligament reconstruction (ACLR) at 6 and 8-week posttests.

ELIGIBILITY:
Inclusion Criteria:

* Have completed all other formal physical therapy
* Are between the ages of 18 and 35
* Underwent an ACLR between 6 and 24 months prior to enrollment.
* Demonstrate underloading during gait (vGRF- impact peak <1.09 x BW)
* Demonstrate clinically relevant-knee symptoms (KOOS-QOL <72)
* Have undergone ACLR surgery

Exclusion Criteria:

* ACLR revision surgery
* A multiple ligament surgery
* A lower extremity fracture
* Knee osteoarthritis
* The participant has a BMI ≥ 36.

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2021-08-05 (Actual); Primary Completion 2022-12-02 (Actual); Study Completion 2022-12-02 (Actual)

PRIMARY OUTCOMES:
Number of participants recruited using different recruitment modes | Baseline (pre-intervention)
  The investigators will record the number of participants who were recruited, the frequency at which they were recruited, and where they were recruited from. Range 0-70. Higher number indicates more completion.
The frequency of participant recruitment using different recruitment modes | Baseline (pre-intervention)
  The investigators will record the number of participants who were recruited, the frequency at which they were recruited, and where they were recruited from. Range 0-70. Higher number indicates more completion.
Percentage of participants who were successfully enrolled | Baseline (pre-intervention)
  The investigators will record the number of participants who were successfully enrolled compared to the total number of participants screened. Range: 0-100. Higher percentage indicates more enrollment.
Percentage of participants retained | After week 4 and after week 8
  Investigators will record the percentage of patients retained at each monthly data capture timepoint.
Reasons for refusal to enroll | Baseline (pre-intervention)
  Investigators will record the reasons participants opt not to enroll in the study to determine whether there is a trend.
Number of subjects who adhered to the intervention | About 2 months
  Percent of subjects who completed the sequence of training sessions and retention sessions. Range: 0-100. Higher percentage indicates more completion

SECONDARY OUTCOMES:
The change in vertical ground reaction force before and after intervention | Up to 2 months
  Participants walked on a dual-belt force-sensing treadmill for 3000 steps while vertical ground reaction forces were collected. This will be collected at Baseline (pre-intervention), Week 6 posttest, and Week 8 posttest. An increase in vertical ground reaction force at weeks 6 and 8 from baseline indicates improved gait mechanics
The change in T1ρ MRI relaxation times before and after intervention | Up to 2 months
  MRI imaging provided cartilage compositions that were used to measure T1ρ relaxation times. The T1ρ MRI relaxation times refer to the proteoglycan density within the tibial and femoral cartilage. This will be collected at Baseline (pre-intervention), Week 6 posttest, and Week 8 posttest. Lower T1rho relaxation times reflects a better outcome.
The change in T1ρ MRI relaxation times in the medial femoral condyle before and after intervention | Up to 2 months
  MRI marker of T1rho relaxation times of medial femoral articular cartilage (i.e proteoglycan density). This will be collected at Baseline (pre-intervention), Week 6 posttest, and Week 8 posttest.
The change in T1ρ MRI relaxation times in the lateral femoral condyle before and after intervention | Up to 2 months
  MRI marker of T1rho relaxation times of lateral femoral articular cartilage (i.e proteoglycan density). This will be collected at Baseline (pre-intervention), Week 6 posttest, and Week 8 posttest.
The change in T1ρ MRI relaxation times in the medial tibial condyle before and after intervention | Up to 2 months
  MRI marker of T1rho relaxation times of medial tibial articular cartilage (i.e proteoglycan density). This will be collected at Baseline (pre-intervention), Week 6 posttest, and Week 8 posttest.
The change in T1ρ MRI relaxation times in the lateral tibial condyle before and after intervention | Up to 2 months
  MRI marker of T1rho relaxation times of lateral tibial articular cartilage (i.e proteoglycan density). This will be collected at Baseline (pre-intervention), Week 6 posttest, and Week 8 posttest.
The change in the Knee Injury and Osteoarthritis Outcome Quality of Life subscale score | Up to 2 months
  Knee injury Osteoarthritis Outcome Score (KOOS) Quality of Life subscale to measure knee-related quality of life at pre-intervention (baseline). This will be collected at Baseline (pre-intervention), Week 6 posttest, and Week 8 posttest. A higher score indicates better knee-related quality of life. Range: 0-100.
The change in the International Knee Documentation Committee Subjective Knee Evaluation form score | Up to 2 months
  The International Knee Documentation Committee (IKDC) Subjective Knee Evaluation form is a 10-item survey that determines patient-reported knee-related function. This will be collected at Baseline (pre-intervention), Week 6 posttest, and Week 8 posttest. A higher score indicates better knee function. Range: 0-100.
The change in the Tegner Activity Scale score | Up to 2 months
  The Tegner Activity Scale (TAS) to quantify activity levels in individuals with ACL injury on an 11-point Likert scale. A higher score indicates a higher level of activity (e.g., a 10 indicates participants compete in professional or collegiate levels of sport on a regular basis while a 0 indicates indicates that participants are unable to complete any sport or recreational activity due to disability). This will be collected at Baseline (pre-intervention), Week 6 posttest, and Week 8 posttest.
The change in the Anterior Cruciate Ligament Return to Sport After Injury Scale score | Up to 2 months
  The Anterior Cruciate Ligament Return to Sport After Injury (ACL-RSI) scale to measure an individual's psychological readiness to return to sport. Range: 0-100 points. A lower score on this questionnaire indicates poorer psychological readiness. This will be collected at Baseline (pre-intervention), Week 6 posttest, and Week 8 posttest.
The change in the Visual, Aural, Reading/Writing, and Kinesthetic Questionnaire score | Up to 2 months
  The Visual, Aural, Reading/Writing, and Kinesthetic (VARK) Questionnaire to quantify a participant's preferred learning styles from four learning styles (Visual, Aural, Reading/Writing, and Kinesthetic). Range: 0-16 for each learning style. Higher scores in one learning style indicates the participant's preferred learning style. This will be collected at Baseline (pre-intervention), Week 6 posttest, and Week 8 posttest.
The change in peak vGRF | Up to 2 months
  Gait biomechanics collected using an eight camera three-dimensional motion analysis system while participants walk on a dual-belt, force-sensing treadmill will be used to quantify peak vGRF. This will be collected at Baseline (pre-intervention), Week 6 posttest, and Week 8 posttest.
The change in peak knee flexion excursion | Up to 2 months
  Gait biomechanics collected using an eight camera three-dimensional motion analysis system while participants walk on a dual-belt, force-sensing treadmill will be used to quantify peak knee flexion excursion. This will be collected at Baseline (pre-intervention), Week 6 posttest, and Week 8 posttest.
The change in peak internal knee extension moment | Up to 2 months
  Gait biomechanics collected using an eight camera three-dimensional motion analysis system while participants walk on a dual-belt, force-sensing treadmill will be used to quantify peak internal knee extension moment. This will be collected at Baseline (pre-intervention), Week 6 posttest, and Week 8 posttest.
The change in joint tissues metabolism by assessing biomarker chemokine (monocyte chemoattractant protein-1 (MCP-1)). | Up to 2 months
  Blood for serum-based biomarker chemokine (monocyte chemoattractant protein-1 (MCP-1)). This will be collected at Baseline (pre-intervention), Week 6 posttest, and Week 8 posttest.
The change in joint tissues metabolism by assessing degenerative matrix metalloproteinase-3 (MMP-3) enzyme. | Up to 2 months
  Blood for serum-based biomarker degenerative matrix metalloproteinase-3 (MMP-3) enzyme. This will be collected at Baseline (pre-intervention), Week 6 posttest, and Week 8 posttest.
The change in joint tissues metabolism by assessing marker of cartilage turnover (cartilage oligomeric matrix protein (COMP)). | Up to 2 months
  Blood for serum-based biomarker marker of cartilage turnover (cartilage oligomeric matrix protein (COMP)). This will be collected at Baseline (pre-intervention), Week 6 posttest, and Week 8 posttest.

CONTACTS AND LOCATIONS:
Overall Officials: Brian Pietrosimone, Principal Investigator — University of North Carolina, Chapel Hill
Locations (1):
- University of North Carolina at Chapel Hill, Chapel Hill, North Carolina, United States

IPD SHARING:
Plan to Share IPD: Yes
Deidentified individual data that supports the results will be shared beginning 9 to 36 months following publication provided the investigator who proposes to use the data has approval from an Institutional Review Board (IRB), Independent Ethics Committee (IEC), or Research Ethics Board (REB), as applicable, and executes a data use/sharing agreement with UNC.
Time Frame: 9 to 36 months
Access Criteria: The investigator who proposes to use the data has approval from an IRB, IEC, or REB, as applicable, and an executed data use/sharing agreement with UNC.